CLINICAL TRIAL: NCT07110961
Title: The Pilot Study of the Utilization of Suggested Immobilization Test (SIT) for Diagnostic Confirmation of Restless Leg Syndrome in Thai Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Jindapa Srikajon, Principal investigator, Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 645/2568(IRB4)
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Restless Leg Syndrome
Keywords: restless leg syndrome; sleep; suggested immobilization test
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Intervention Model Description: All participants will undergo a suggested immobilization test on the same day of the sleep test appointment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical diagnosed restless leg syndrome (Experimental): Participants with appointment of sleep test and clinical diagnosed restless leg syndrome according to International Restless Legs Syndrome Study Group (IRLSSG) are reruited and undergo a suggested immobilization test before the standard polysomnographic study.
  Interventions: Procedure: A suggested immobilization test (SIT)

INTERVENTIONS:
Procedure: A suggested immobilization test (SIT) — The Suggested Immobilization Test (SIT) is a provocative test. RLS symptoms (urge to move the leg and leg paresthesia) are primarily observed during wakefulness, especially at rest, in the evening, and/or during the night. During the test, the patient remains in a bed (or a reclining chair), at a 45° angle with legs outstretched. Originally, the SIT only quantified leg motor activity. Since 2002, it also includes the assessment of leg discomfort, which is estimated by the patient every 5 min, on a 100-mm horizontal visual analogue scale. Leg movements are quantified using surface electromyography (EMG) from bilateral anterior tibialis muscles. Using these pathological thresholds, the clinical RLS/WED diagnosis is correctly predicted in 88% of subjects with a sensitivity of 82% and a specificity of 100%.

SUMMARY:
Restless leg syndrome (RLS) is not uncommon and can also affect people's health and quality of life. Mainly, RLS is diagnosed based on clinical criteria subjectively. Sometimes it is difficult to differentiate between RLS and mimickers, especially in patients with comorbidities such as diabetes or parkinson's disease. We believe that using objective tests would facilitate accuracy in RLS diagnosis, which leads to proper management of patients.

DETAILED DESCRIPTION:
Restless legs syndrome (RLS) represents disturbing symptoms in the lower limbs that lead to the urge to move, occurring in rest periods. Movements can partially or completely relieve these abnormal feelings. In 2014, the International RLS Study Group (IRLSSG) established five mandatory criteria for the diagnosis of RLS1.

IRLSSG essential diagnostic criteria for RLS (all must be met):

* An urge to move the legs, usually but not always accompanied by, or felt to be caused by, uncomfortable and unpleasant sensations in the legs
* The urge to move the legs and any accompanying unpleasant sensations begin or worsen during periods of rest or inactivity, such as lying down or sitting
* The urge to move the legs and any accompanying unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues
* The urge to move the legs and any accompanying unpleasant sensations during rest or inactivity only occur or are worse in the evening or night than during the day.
* The occurrence of the above features is not solely accounted for as symptoms primary to another medical or a behavioral condition (e.g., myalgia, venous stasis, leg edema, arthritis, leg cramps, positional discomfort, habitual foot tapping) In the general population, a prevalence of RLS was reported up to 10%2. The prevalence of RLS varies considerably depending on the methods of diagnosis, country, sex, age, and comorbidity burden, which impedes comparisons between studies3. Generally, the prevalence of RLS is relatively low, approximately 1% in Asian populations4-6. In contrast, the prevalence of RLS is considerably higher, ranging from 5% to 10% in Europe and North America7. A cross-sectional nationwide survey of 6,509 Korean adults aged 18-64, using criteria established by the International RLS Study Group (IRLSSG) to define RLS, found a prevalence of 0.9% (0.6% in men and 1.3% in women)5. There was only one study focusing on the prevalence of RLS in Thailand, in which the prevalence of RLS in Thai Parkinson's patients was only 1.6%8.

The nonpharmacologic treatment of RLS includes stretching, heating, or cooling the extremities (e.g., a warm bath), and avoiding alcohol and caffeine. However, the U.S. Food and Drug Administration (FDA) has not approved physical devices such as compression stockings, heating and vibrating pads, and foot pressure wraps for the treatment of RLS9.

Pharmacologic treatment: The latest clinical practice guideline (CPG) updates the 2024 American Academy of Sleep Medicine (AASM) practice parameters and offers new recommendations for treating RLS in adult patients. The primary change in these recommendations is the inclusion of alpha-2-delta ligands (gabapentin, gabapentin enacarbil, and pregabalin) in the 'strong recommendation' category, along with a transition from the use of dopamine agonists to a 'conditional recommendation' in order to mitigate side effects such as augmentation and impulse control disorders 10.

Patients with RLS experience significant adverse effects on work performance, quality of life, cognition, and health11,12. A survey study conducted in the United States that examined the disease burden of primary RLS found that work productivity is diminished by approximately 20%, which equates to about one day per 40-hour work week for individuals with moderate to severe RLS. The mean EQ-5D health utility score indicated a significantly lower health status compared to the healthy control group. Additionally, RLS negatively impacts sleep quality, with 60-70% of patients reporting poor sleep11. RLS not only causes impaired quality of life but also possibly leads to cardiovascular consequences. RLS was associated with statistically significantly less future cardiovascular risk in RLS patients with treatment than in those without treatment13.

The diagnosis of RLS is primarily based on a clinical history of an urge to move the limbs that worsens when at rest, improves with movement, and is more prominent in the evening or at night. These four criteria have a positive predictive value (PPV) of 76% when an expert interview is used as the gold standard. Carefully distinguishing RLS from leg cramps or positional discomfort increases the specificity of the four criteria from 84% to 94%14. However, some RLS mimics, such as nocturnal leg cramps or neuropathy, still cannot be addressed solely by clinical history or basic RLS screening instruments. Consequently, there should be standardized objective tests for RLS beyond clinical diagnosis.

The Suggested Immobilization Test (SIT) is a provocative test. RLS symptoms (urge to move the leg and leg paresthesia) are primarily observed during wakefulness, especially at rest, in the evening, and/or during the night. During the test, the patient remains in a bed (or a reclining chair), at a 45° angle with legs outstretched. Originally, the SIT only quantified leg motor activity. Since 2002, it also includes the assessment of leg discomfort, which is estimated by the patient every 5 min, on a 100-mm horizontal visual analogue scale. Leg movements are quantified using surface electromyography (EMG) from bilateral anterior tibialis muscles. Using these pathological thresholds, the clinical RLS/WED diagnosis is correctly predicted in 88% of subjects with a sensitivity of 82% and a specificity of 100%15,16.

It was not only used for diagnosis but also for measuring the severity of symptoms. Patients with severe RLS show more leg movements during the SIT than those with moderate or mild RLS. Additionally, it can help differentiate RLS mimics, which can be challenging with only a clinical diagnosis, as mentioned above. Moreover, it would benefit special populations, especially those with Parkinson's disease or Multiple sclerosis, who have some symptoms that could confound the diagnosis of restless leg syndrome17,18. The low cost and the ability to repeat the tests multiple times throughout the day are the two main advantages of SIT. It can also be done on the same day as a routine sleep test.

To the best of investigator's knowledge, this is the first pilot study of SIT for confirmation of restless leg syndrome in the Thai population. Early diagnosis with a high-accuracy test would lead to appropriate treatment planning and better outcomes in Thai RLS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were appointed for an in-lab polysomnographic study and fit the clinical diagnosis criteria for restless leg syndrome based on International Restless Legs Syndrome Study Group (IRLSSG)

Exclusion Criteria:

* Patient with physical limitations including stroke, dementia or hearing impairment
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between clinical diagnosis based on criteria and results from a suggested immobilization test | During intervention
  Between-group and correlation analyses between categorical and continuous data were corrected using Spearman's rank correlation.

SECONDARY OUTCOMES:
Occurence of advense events from a suggested immobilization test | During intervention
  discomfort or any unconfotable feeling during the test will be recorded.

IPD SHARING:
Plan to Share IPD: Undecided
Still deciding

REFERENCES:
- See also: Related Info — https://www.irlssg.org